CLINICAL TRIAL: NCT02006329
Title: Treatment of Non Alcoholic Fatty Liver Disease With Lifestyle Modification and Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Assy Nimer, MD, Ziv Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0089-13-ziv
Record Dates: First submitted 2013-11-27; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: NAFLD; Accupuncture
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Acupuncture Therapy

ARMS (2):
- Intervention group - dietary consultation - Medit (Experimental)
  Interventions: Device: acupuncture
- Control group - dietary consultation - Mediterranean diet (No Intervention)

INTERVENTIONS:
Device: acupuncture
  Arms: Intervention group - dietary consultation - Medit

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of liver dysfunction worldwide. NAFLD may progress to nonalcoholic steatohepatitis (NASH) and in turn to cirrhosis. To date, the detailed pathogenic mechanism of NAFLD including steatosis and NASH is not fully characterized, although it is regarded as a hepatic manifestation of the metabolic syndrome, sometimes it occurs in the absence of a metabolic syndrome. Based on conventional models of "two-hit" and "multi- hit" hypothesis of NAFLD, the dysregulated lipid metabolism and insulin resistance are considered as the "first hit" of the liver and the following "second hit" or "multi-hit" likely involves oxidative stress, lipid peroxidation, increased inflammatory responses, induced hepatic fibrosis and apoptosis. This emphasizes the multi-factorial pathogenesis of NAFLD and the necessity to treat NAFLD with diabetes-like and multimodal strategy. Several changes in dietary intake have occurred in the past few years, including increased energy intake (24%), and increases in added sugars, flour and cereal products, fruit, added fats and total fat intake. The increasing prevalence of NAFLD is probably directly affected by the contemporary epidemics of obesity, unhealthy dietary pattern, and sedentary lifestyle. Currently, there are two major categories of NAFLD therapy: lifestyle interventions and pharmaceutical therapies, lifestyle interventions in terms of diet and physical activity are regarded as safe and effective, while pharmaceutical interventions showed limited efficacy with unknown safety in the long term ,therefore, the first line of treatment is lifestyle modification. Although lifestyle intervention dose positively affects NAFLD, it has limitations. Patients adherence to dietary intervention is 50%, while those who do adhere, find it difficult to maintain after 12 months. ). Mediterranean diet has been shown to be effective in reducing NAFLD, liver steatosis and improve insulin sensitivity. Acupuncture has been found as an effective treatment for improving quality of life in various medical conditions , including hepatitis . Acupuncture combined with life style intervention has been found effective in the treatment of obesity, metabolic syndrome in terms of weight, lipid regulation, glucose levels and various markers of inflammation. Acupuncture's effect on NAFLD has yet to be studied.

We suggest that acupuncture combined with life style intervention can be an effective treatment for NAFLD.

ELIGIBILITY:
Inclusion Criteria:

Above 18 years old No known metabolic pathology NAFLD diagnosis

Exclusion Criteria:

Known metabolic pathology Psychiatric diagnosis Auto immune disease Known Diabetes Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Fibroscan test | 3 months after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel, Israel